CLINICAL TRIAL: NCT01735500
Title: Rise of hscTnT After Elective Coronary Angiography Without Coronary Intervention
Brief Title: hsTnT After Elective Coronary Angiography
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Haitham Abu Sharar, Dr. med., University Hospital Heidelberg
Other Study IDs: hsTnT Elective CAG
Record Dates: First submitted 2012-11-24; First posted 2012-11-28 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease
Keywords: Prei-procedural; Elevation; cardia Troponin T; in stable; unknown
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- CAG without PCI
- CAG with PCI

SUMMARY:
A prospective Study, aiming to understand and analyse the key role of the novel High Sensitivity Troponin T (hsTnT) within a group of patients undergoing an uncomplicated coronary angiography without receiving any additional intervention. The peri-procedural elevation of the hsTnT indicates some other factors being responsible for the elevation of the hsTnT in absence of an acute coronary syndrome, such as physiological components or micro-injuries. A one year follow-up has been collected.

ELIGIBILITY:
Inclusion Criteria:

- Stable or unknown CAD

Exclusion Criteria:

- Acute Coronary Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with stable or unknown CAD undergoing CAG with/or without PCI. Patients receiving additional examination, such as biopsy, Ablation or any other procedure that could lead to myocardial injury resulting in elevation of the cardiac Troponin are being excluded, as well as Patients with acute coronary syndrome.
Sampling Method: Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | Up to 12 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giannitsis, Prof. Dr. med., Principal Investigator — Department of Cardiology, University Hospital of Heidelberg
Locations (1):
- Department of Cardiology - University Hospital of Heidelberg, Heidelberg, Germany